CLINICAL TRIAL: NCT05178888
Title: A Phase 1/1b Trial of MRTX849 in Combination With Palbociclib in Patients With Advanced Solid Tumors With KRAS G12C Mutation
Brief Title: Adagrasib in Combination With Palbociclib in Patients With Advanced Solid Tumors (KRYSTAL-16)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0018; CA239-0018 (Other: Bristol-Myers Squibb Protocol ID); 849-016 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — adagrasib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation of MRTX849 and palbociclib to determine maximum tolerated dose in combination.
  Interventions: Drug: MRTX849; Drug: Palbociclib
- Dose Expansion (Experimental): Expansion cohorts may be implemented to ensure sufficient safety experience, pharmacokinetic data and early evidence of clinical activity of MRTX in combination with palbociclib.
  Interventions: Drug: MRTX849; Drug: Palbociclib

INTERVENTIONS:
Drug: MRTX849 — KRAS G12C inhibitor
  Other Names: KRAS G12C; adagrasib
Drug: Palbociclib — CDK 4 and 6 inhibitor
  Other Names: IBRANCE

SUMMARY:
This study will evaluate the safety and clinical activity of MRTX849 (adagrasib) in combination with palbociclib in patients with advanced solid tumor malignancies with KRAS G12C mutation.

DETAILED DESCRIPTION:
This study will evaluate the pharmacokinetics and preliminary clinical activity of MRTX849 (adagrasib) in combination with palbociclib in patients with advanced solid tumor malignancies with KRAS G12C mutation. MRTX849 is an orally available small molecule inhibitor of KRAS G12C and palbociclib is a small molecule inhibitor of CDK 4 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy with KRAS G12C mutation
* Unresectable or metastatic disease.
* No available treatment with curative intent
* Adequate organ function

Exclusion Criteria:

* History of significant toxicity on prior KRAS G12C or CDK4/6 inhibitor therapies
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter the absorption of study treatment or result in an inability to swallow
* Other active cancer
* Cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Characterize the number of patients with treatment emergent adverse events of the combination regimen in patients with advanced solid tumor malignancies with KRAS G12C mutation. | 24 months
  Number of participants with treatment emergent adverse events
Evaluate Pharmacokinetics of the combination regimen | 24 months
  Plasma concentration
Establish Maximum Tolerated Dose | 24 months
  Number of patients with dose limiting toxicity
Evaluate preliminary clinical activity of the combination regimen | 24 months
  Objective response rate in accordance with Response Evaluation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution - 804, Orlando, Florida
  - Local Institution - 803, Nashville, Tennessee
  - Local Institution - 802, Houston, Texas
  - Local Institution - 801, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com